CLINICAL TRIAL: NCT01560975
Title: A Prospective, Explorative, Open Label Study to Assess the 24-hour Intraocular Pressure Fluctuation Profile Recorded With SENSIMED Triggerfish® in Patients With Moderate to Severe Obstructive Sleep Apnea Syndrome Using Continuous Positive Airway Pressure With or Without Primary Open Angle Glaucoma
Brief Title: IOP Fluctuations in Patients With Sleep Apnea With or Without Primary Open Angle Glaucoma Using Positive Airway Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1108
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Sleep Apnea, Obstructive; Primary Open-angle Glaucoma
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sensimed Triggerfish (Experimental)
  Interventions: Device: SENSIMED Triggerfish®

INTERVENTIONS:
Device: SENSIMED Triggerfish® — Portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours

SUMMARY:
Sleep apnea is characterized by repetitive episodes of decreased or interrupted airflow in the upper airways during sleep. Obstructive sleep apnea syndrome (OSAS) is the most common sleep-related breathing disorder and is characterized by repeated partial or complete upper airway collapse, gasping episodes, daytime sleepiness and fatigue. Once suspected, the diagnosis is made on the basis of anamnesis and a polysomnography (PSG) using the so-called respiratory disturbance index (RDI) to grade OSAS. Standard therapy consists of continuous positive airway pressure (CPAP) during sleep to prevent upper airway collapse. The association between OSAS and glaucoma has been extensively studied, although a few reports have been non-confirmatory. OSAS has been associated with reduced ocular blood flow, leading to hypoxia and hypercapnia, and as such, may represent a risk factor for glaucomatous optic neuropathy. OSAS has also been related to loss of nycthemeral rhythm of intraocular pressure (IOP). In addition, CPAP has been reported to increase IOP when used during nighttime.

The purpose of this study is to investigate how IOP varies in time, particularly during sleep in OSAS patients with or without glaucoma, and if the IOP variations are associated with the use of CPAP. IOP fluctuations will be monitored with SENSIMED Triggerfish®, a portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of moderate to severe OSAS, determined by a RDI > 15 on PSG
* Patient has either POAG with controlled IOP or no glaucoma. Five of each will included in the study
* Patients under CPAP therapy
* Aged ≥ 18 years, of either sex
* Not more than 4 diopters spherical equivalent on the study eye
* Not more than 2 diopters cylinder equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Sleep disorders other than OSAS
* Use of sleep medication
* Patients with history of intraocular surgery (including laser therapy) within the last 3 months
* Corneal or conjunctival abnormality hindering contact lens adaptation
* Severe dry eye syndrome
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 30 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — The New York Eye and Ear infirmary
Locations (1):
- The New York Eye and Ear Infirmary, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensimed Triggerfish
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sensimed Triggerfish
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between IOP Fluctuation Pattern With or Without CPAP Therapy in Patients With Moderate to Severe OSAS With or Without POAG
Description: 24-hour IOP fluctuation pattern recorded using Triggerfish in patients with moderate to severe OSAS.
  * using CPAP in patients with or without POAG
  * not using CPAP in patients with or without POAG
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mVEq/h
Groups:
- POAG/CPAP: POAG patients with CPAP therapy
- noPOAG/CPAP: Subjects with CPAP
Arm/Group | POAG/CPAP | noPOAG/CPAP
Number analyzed (Participants) | 4 | 4
mVEq/h | 44.4 (34.8) | 42.2 (40.7)

2. Secondary Outcome: Relationship Between the 24-hour IOP Fluctuation Patterns and Physiologic Parameters
Description: Heart rate and ocular pulsation rate during sleep:
  * using CPAP in patients with or without POAG
  * not using CPAP in patients with or without POAG
Time Frame: 24-hours
Measure: Mean (Standard Deviation); unit: Correlation
Groups:
- noPOAG/CPAP: no POAG patients with CPAP therapy
- POAG/no CPAP: POAG patients without CPAP therapy
- noPOAG/ no CPAP: No POAG patients without CPAP therapy
Arm/Group | POAG/CPAP | noPOAG/CPAP | POAG/no CPAP | noPOAG/ no CPAP
Number analyzed (Participants) | 4 | 4 | 4 | 4
Correlation | 0.36 (0.4) | 0.92 (0.03) | 0.47 (0.33) | 0.42 (0.20)

3. Secondary Outcome: Effect After CPAP Removal on the IOP Pattern
Description: IOP pattern immediately after CPAP removal upon waking in patients with or without POAG
Time Frame: 30 min
Measure: Mean (Standard Deviation); unit: mvEq
Arm/Group | POAG/CPAP | noPOAG/CPAP | POAG/no CPAP | noPOAG/ no CPAP
Number analyzed (Participants) | 4 | 4 | 4 | 4
mvEq | -2.6 (54) | -25.4 (69.1) | -40.4 (89.2) | -50.3 (91.2)

ADVERSE EVENTS:
Arm/Group | Sensimed Triggerfish
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No